CLINICAL TRIAL: NCT00450203
Title: A Randomised Phase II/III Trial of Peri-Operative Chemotherapy With or Without Bevacizumab in Operable Oesophagogastric Adenocarcinoma and A Feasibility Study Evaluating Lapatinib in HER-2 Positive Oesophagogastric Adenocarcinomas and (in Selected Centres) MRI and PET/CT Sub-studies
Brief Title: Chemotherapy With or Without Bevacizumab or Lapatinib to Treat Operable Oesophagogastric Cancer
Acronym: ST03
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Professor David Cunningham (Other Government)
Collaborators: Cancer Research UK (Other); Roche Pharma AG (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Professor David Cunningham, ST03 Chief Investigator, Professor David Cunningham, Medical Research Council
Organization: Medical Research Council (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000536013; MRC-ST03 (Other: MRC); EU-20710; ISRCTN46020948 (Other: ISRCTN); 2006-000811-12 (EudraCT Number); 00316/0221/001 (Other: CTA)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Oesophagogastric Cancer
Keywords: adenocarcinoma of the stomach; adenocarcinoma of the gastro oesophageal junction; adenocarcinoma of the lower oesophagus
MeSH Terms: interventions — Bevacizumab; Capecitabine; Cisplatin; Epirubicin; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ECX + Bevacizumab (Experimental): ECX + Bevacizumab
  Interventions: Biological: bevacizumab; Drug: capecitabine; Drug: cisplatin; Drug: Epirubicin; Procedure: adjuvant therapy; Procedure: conventional surgery; Procedure: neoadjuvant therapy
- Epirubicin, Cisplatin and Capecitabine (Active Comparator): ECX chemotherapy
  Interventions: Drug: capecitabine; Drug: cisplatin; Drug: Epirubicin; Procedure: adjuvant therapy; Procedure: conventional surgery; Procedure: neoadjuvant therapy
- ECX + Lapatinib (Experimental): ECX + Lapatinib
  Interventions: Drug: capecitabine; Drug: cisplatin; Drug: Epirubicin; Procedure: adjuvant therapy; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Drug: Lapatinib

INTERVENTIONS:
Biological: bevacizumab — 7.5mg/kg IV Day 1 of each 21 cycle of chemotherapy (6 cycles) plus day 1 of each maintenance dose every 21 days for 6 doses.
  Arms: ECX + Bevacizumab
Drug: capecitabine — dose banded as based on patient BSA. Oral dose given twice a day during each 21 day cycle of chemotherapy (6 cycles in total)
Drug: cisplatin — 60mg/m2 IV day one of each 21 day cycle of chemotherapy (6 cycles in total)
Drug: Epirubicin — 50mg/m2 IV day one of each 21 day cycle of chemotherapy (6 cycles in total)
Procedure: adjuvant therapy — 3 cycles of ECX chemotherapy post operatively
Procedure: conventional surgery — Surgery undertaken after 3 cycles of pre-operative chemotherapy. Followed by 3 cycles of chemotherapy.
Procedure: neoadjuvant therapy — 3 cycles of pre-operative ECX chemotherapy.
Drug: Lapatinib — 1250mg/day Day 1-21 of each cycle of chemotherapy (6 cycles) plus day 1-21 of each maintenance course every 21 days for 6 doses.
  Other Names: Tyverb
  Arms: ECX + Lapatinib

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as epirubicin, cisplatin, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, and small molecule tyrosine kinase inhibitors, such as lapatinib, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Lapatinib targets a specific growth receptor, HER-2. Chemotherapy together with bevacizumab or lapatinib, in HER-2 positive tumours, may kill more tumor cells.

PURPOSE: This randomized phase II/III trial is studying the side effects and how well giving combination chemotherapy together with bevacizumab works compared with combination chemotherapy alone in treating patients with previously untreated stomach cancer, gastroesophageal junction cancer or lower oesophageal cancer that can be removed by surgery. The feasibility study is studying the safety of adding lapatinib to chemotherapy in patients with HER-2 positive previously untreated stomach cancer, gastroesophageal junction cancer or lower oesophageal cancer that can be removed by surgery. The feasibility study will also assess the feasibility of timely HER-2 testing and estimate the HER-2 positivity rate in this patient population.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the safety and efficacy of neoadjuvant and adjuvant chemotherapy comprising epirubicin hydrochloride, cisplatin, and capecitabine with or without bevacizumab in patients with previously untreated, resectable gastric, gastroesophageal junction or lower oesophageal cancer.
* Assess the safety of neoadjuvant and adjuvant chemotherapy comprising epirubicin hydrochloride, cisplatin, and capecitabine with or without lapatinib in patients with HER-2 positive previously untreated, resectable gastric, gastroesophageal junction or lower oesophageal cancer.

OUTLINE: This is a multicenter, randomized, open-label, controlled study. Patients are randomized to 1 of 4 treatment arms.

* Arm I and II: Patients receive epirubicin hydrochloride IV and cisplatin IV over 4 hours on day 1 and capecitabine orally twice daily on days 1-21. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo surgery 5-6 weeks after completion of chemotherapy. Patients then receive 3 additional courses of chemotherapy beginning 6-10 weeks after surgery.

* Arm II: Patients receive bevacizumab IV over 30-90 minutes, epirubicin hydrochloride IV, and cisplatin IV over 4 hours on day 1 and capecitabine orally twice daily on days 1-21. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo surgery 5-8 weeks after completion of chemotherapy. Patients then receive 3 additional courses of chemotherapy and bevacizumab beginning 6-10 weeks after surgery. Patients then receive maintenance therapy comprising bevacizumab IV over 30-90 minutes on day 1. Maintenance therapy repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

* Arm IV: Patients receive lapatinib orally once daily, epirubicin hydrochloride IV, and cisplatin IV over 4 hours on day 1 and capecitabine orally twice daily on days 1-21. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo surgery 5-8 weeks after completion of chemotherapy. Patients then receive 3 additional courses of chemotherapy and lapatinib beginning 6-10 weeks after surgery. Patients then receive maintenance therapy comprising lapatinib orally once daily on days 1-21. Maintenance therapy repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, during treatment, and during the follow-up period.

After completion of study treatment, patients are followed at 9, 18, and 27 weeks after the start of course 4, 1 year post surgery, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 1063 patients were recruited to the bevacizumab comparison of the study (now closed to recruitment) and 40 patients with HER-2 positive tumours will be recruited into the ST03 feasibility study.

ELIGIBILITY:
This is a combined eligibility criteria for both bevacizumab comparison and the lapatinib feasibility study. Please note the bevacizumab comparison closed to recruitment on 28th March 2014.

DISEASE CHARACTERISTICS:

* Histologically confirmed gastric or type I, II or III gastroesophageal junction adenocarcinoma or lower oesophageal

Gastric and Type III junctional tumours should be Stage Ib (T1 N1, T2a/b N0), II, III or stage IV (T4 N1 or N2) with no evidence of distant metastases (M0)

Lower oesophageal and Type I and II junctional tumours should be Stage II to Stage IVa (T1 N1, T2 N1, T3 N0-1, but not T2N0). T4 (N0 or N1) tumours are also eligible providing that they involve only the crura OR invade only the mediastinal pleura. Patients with nodal disease affecting the origin of the left gastric and splenic artery or coeliac axis (staged as M1a) are also eligible.

* Resectable disease
* Previously untreated disease

PATIENT CHARACTERISTICS:

* WHO performance status 0 or 1
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL (can be post transfusion)
* WBC ≥ 3,000/mm^3
* Glomerular filtration rate ≥ 60 mL/min
* Proteinuria ≤ 1 g by 24-hour urine collection
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 3 times ULN (in the absence of liver metastases)
* INR ≤ 1.5
* PTT ≤ 1.5 times ULN
* FEV_1 ≥ 1.5 L
* Cardiac ejection fraction ≥ 50% by MUGA scan or echocardiogram
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must be fit enough to receive protocol treatment
* No other malignancies within the past 5 years except for curatively treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix
* No prior or concurrent significant medical conditions, including any of the following:

  * Cerebrovascular disease (including transient ischemic attack and stroke) within the past year
  * Cardiovascular disease, including the following:

    * Myocardial infarction within the past year
    * Uncontrolled hypertension while receiving chronic medication
    * Unstable angina
    * New York Heart Association class II-IV congestive heart failure
    * Serious cardiac arrhythmia requiring medication
  * Major trauma within the past 28 days
  * Serious nonhealing wound, ulcer, or bone fracture
  * Evidence of bleeding diathesis or coagulopathy
  * Recent history of any active gastrointestinal inflammatory condition (e.g., peptic ulcer disease, diverticulitis, or inflammatory bowel disease)

    * If patients have a known diagnosis of any of the above, evidence of disease control is required by negative endoscopy within the past 28 days
* No severe tinnitus
* No lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication
* No known peripheral neuropathy ≥ 1 (absence of deep tendon reflexes as the sole neurological abnormality does not render the patient ineligible)
* No known dihydropyrimidine dehydrogenase deficiency
* No history of interstitial lung disease or radiological evidence of lung fibrosis
* No known allergy to any of the following:

  * Chinese hamster ovary cell proteins
  * Other recombinant human or humanized antibodies
  * Any excipients of bevacizumab formulation or platinum compounds
  * Any other components of the study drugs

Due to an increase in perforations associated with self-expandable metal stents in patients with colorectal cancer receiving bevacizumab, patients with an oesophageal or gastric stent (metal or biodegradable) in situ are ineligible for the study.

PRIOR CONCURRENT THERAPY:

* No prior anthracycline
* More than 28 days since prior major surgery or open biopsy
* More than 10 days since prior thrombolytic therapy
* No concurrent thrombolytic therapy
* No concurrent dipyridamole
* No concurrent capecitabine or sorivudine (or sorivudine analogues [e.g., brivudine])
* No chronic, daily high-dose acetylsalicylic acid (> 325 mg/day) or nonsteroidal anti-inflammatory drugs
* No chronic corticosteroids (≥ 10 mg/day methylprednisolone equivalent)

  * Inhaled steroids allowed
* No other concurrent cytotoxic agents
* No other concurrent investigational drugs
* No concurrent radiotherapy
* Low molecular weight heparin allowed
* More than 7 days since prior CYP3A4 inhibitor therapy
* More than 14 days since prior CYP3A4 inducer therapy
* More than 6 months since prior amiodarone therapy
* More than 14 days since prior St John's Wort, modafinil, ginkgo biloba, kava, grape seed, valerian, ginseng, echinacea and evening primrose oil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1103 (Estimated)
Dates: Start 2007-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Safety | at the end of phase II and phase III
Efficacy | end of trial
Overall survival | end of trial

SECONDARY OUTCOMES:
Feasibility | end of trial
Treatment-related morbidity | end of trial
Response rates to pre-operative treatment | at phase II review and at end of trial
Surgical resection rates | end of trial
Disease-free survival | end of trial
Quality of life | end of trial
Cost-effectiveness | end of trial
HER-2 Positivity Rate | End of trial
Feasibility of centralised HER-2 testing | After 60 patients tested and then after 110 patients tested and then at end of trial

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, MD, Study Chair — Royal Marsden NHS Foundation Trust
Locations (41):
- United Kingdom (41):
  - Royal Bournemouth Hospital, Bournemouth, England
  - Bradford Royal Infirmary, Bradford, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Cumberland Infirmary, Carlisle, England
  - Doncaster Royal Infirmary, Doncaster, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Lincoln County Hospital, Lincoln, England
  - Aintree University Hospital, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - St. George's Hospital, London, England
  - St. Mary's Hospital, London, England
  - Mid Kent Oncology Centre at Maidstone Hospital, Maidstone, England
  - Christie Hospital, Manchester, England
  - Clatterbridge Centre for Oncology, Merseyside, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Derriford Hospital, Plymouth, England
  - Dorset Cancer Centre, Poole Dorset, England
  - Berkshire Cancer Centre at Royal Berkshire Hospital, Reading, England
  - Rochdale Infirmary, Rochdale, England
  - Salisbury District Hospital, Salisbury, England
  - Wexham Park Hospital, Slough, Berkshire, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Basingstoke and North Hampshire Hospital, Basingstoke
  - Birmingham Heartlands Hospital, Birmingham
  - Castle Hill Hospital, Cottingham
  - University Hospitals Coventry and Warwickshire, Coventry
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Norfolk and Norwich University Hospital, Norwich
  - Churchill Hospital, Oxford
  - Queens Hospital, Romford
  - Weston Park, Sheffield
  - Great Western Hospital, Swindon
  - Musgrove Park Hospital, Taunton

REFERENCES:
- [Result] Okines AF, Langley RE, Thompson LC, Stenning SP, Stevenson L, Falk S, Seymour M, Coxon F, Middleton GW, Smith D, Evans L, Slater S, Waters J, Ford D, Hall M, Iveson TJ, Petty RD, Plummer C, Allum WH, Blazeby JM, Griffin M, Cunningham D. Bevacizumab with peri-operative epirubicin, cisplatin and capecitabine (ECX) in localised gastro-oesophageal adenocarcinoma: a safety report. Ann Oncol. 2013 Mar;24(3):702-9. doi: 10.1093/annonc/mds533. Epub 2012 Oct 28. PMID 23108952
- [Derived] Allum WH, Smyth EC, Blazeby JM, Grabsch HI, Griffin SM, Rowley S, Cafferty FH, Langley RE, Cunningham D. Quality assurance of surgery in the randomized ST03 trial of perioperative chemotherapy in carcinoma of the stomach and gastro-oesophageal junction. Br J Surg. 2019 Aug;106(9):1204-1215. doi: 10.1002/bjs.11184. Epub 2019 Jul 3. PMID 31268180
- [Derived] Cunningham D, Stenning SP, Smyth EC, Okines AF, Allum WH, Rowley S, Stevenson L, Grabsch HI, Alderson D, Crosby T, Griffin SM, Mansoor W, Coxon FY, Falk SJ, Darby S, Sumpter KA, Blazeby JM, Langley RE. Peri-operative chemotherapy with or without bevacizumab in operable oesophagogastric adenocarcinoma (UK Medical Research Council ST03): primary analysis results of a multicentre, open-label, randomised phase 2-3 trial. Lancet Oncol. 2017 Mar;18(3):357-370. doi: 10.1016/S1470-2045(17)30043-8. Epub 2017 Feb 3. PMID 28163000
- See also: Medical Research Council ST03 Clinical Trial Page — http://www.ctu.mrc.ac.uk/research_areas/study_details.aspx?s=33